CLINICAL TRIAL: NCT04973774
Title: A Multi-center Prospective Study of Branch Atheromatous Disease in China
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Bin Peng, Professor, Peking Union Medical College Hospital
Other Study IDs: BADstudy
Record Dates: First submitted 2021-07-17; First posted 2021-07-22 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-07

CONDITIONS: Cerebral Infarction; Disease; Magnetic Resonance Imaging
Keywords: branch atheromatous disease; prospective; tirofiban; antiplatelet; prognosis; Lenticulostriate artery; HRMRI; 3TVWI
MeSH Terms: conditions — Cerebral Infarction; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Branch atheromatous disease (BAD), is regarded as one of the important etiologies for acute isolated subcortical infarction, especially in Asian population. However, due to the fact that the existing imaging techniques cannot depict small vessel changes, the clinical diagnosis, therapy and research of BAD are facing challenges. We have started a multi-center prospective observational study of BAD in China, aiming at establishing a large-sample clinical-radiological cohort of BAD, analyzing predictors for functional outcome, and exploring the efficacy of tirofiban on BAD. A standardized Case Report Form (and eCRF on website) is used to collect baseline and follow-up information on epidemiological, clinical, radiological（MRI, SWI, MRA, HRMRI,3TVWI）and blood test. The primary outcome was mRS on 90 days with blind evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. Age:18-80years
2. Acute cerebral infarction:if the clinical manifestations are TIA, new infarct lesions should be found on DWI at the same time.
3. The time from onset to enrollment is less than 72 hours. If the onset time was unknown, the time of last known free of new ischemic symptoms to enrollment is less than 72h.
4. Meet the following radiological criterial： 1) DWI infarct: single (isolated) deep (subcortical) infarct. 2) The culprit vessels are the lenticulostriate artery or the para-pontine median artery, and the infarct lesion on DWI conforms to one of the following characteri stics(A/B): A. Lenticulostriate artery: ① "comma-like" infarct lesions with "fan-shaped" extension from bottom to top in the coronary position; OR ② ≥3 layers (layer thickness 5-7 mm) on axial DWI images of the head; B. Para-pontine median artery: the infarct lesion extends from the deep pons to the ventral pons on the axial DWI of the head.

3) No ≥50% stenosis on the parent artery of the criminal vessel (i.e. corresponding basilar or middle cerebral artery) (confirmed by MRA or CTA or DSA).

5.Signed informed consent by the patient or legally authorised representatives

Exclusion Criteria:

1. Intracranial hemorrhagic diseases, vascular malformations, aneurysms, brain abscesses, malignant space occupying lesions or other non-ischemic intracranial lesions observed by baseline head CT and MRI, MRA/CTA/DSA;
2. There was ≥50% stenosis of extracranial vessels with ipsally serial relationship
3. Cardiogenic embolism: atrial fibrillation, myocardial infarction, valvular heart disease, dilated cardiomyopathy, infective endocarditis, atrioventricular block disease, heart rate less than 50 beats /min
4. Have received or plan to receive acute endovascular treatment after onset of the disease
5. stroke caused by other clear causes, such as moyamoya disease, arterial dissection, vasculitis, etc
6. mRS score prior to the onset of the disease was ≥2 points
7. Known malignant tumor
8. Life expectancy ≤6 months
9. Can not tolerate 3T MRI examination
10. Pregnant or lactating women
11. Participation in another clinical within 3 months before enrollment, or taking part in another ongoing study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population will include all acute ischemic stroke patients meeting the inclusion and exclusion criteria in all centers of our study.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-05-31 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
modified ranking score | 90 days
  modified ranking score on 90 days, range:0-6scores; higher score means worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Bin Peng, Phd,MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Shengde li, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided